CLINICAL TRIAL: NCT02864901
Title: A Double-Blind, Randomized, Placebo Controlled, Clinical Trial of an Antiplaque Chewing Gum (30 mg) - Phase 2 Proof of Concept in a Generally Healthy Patient Population
Brief Title: Is an Antiplaque Chewing Gum (30 mg) Able to Reduce Dental Plaque in a Healthy Population?
Acronym: APCG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: S-16-10
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Plaque Regrowth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- KSL-W 30 mg (Experimental): 3 times per day over 4 treatment days
  Interventions: Drug: KSL-W
- Chewing Gum Placebo (Placebo Comparator): 3 times per day over 4 treatment days
  Interventions: Drug: KSL-W

INTERVENTIONS:
Drug: KSL-W — Antimicrobial KSL-W Plaque reducing chewing gum
  Other Names: Antimicrobial decapeptide KSL-W

SUMMARY:
The Safety, efficacy and tolerability of an Antimicrobial Chewing Gum Formulation in Reducing Dental Plaque

DETAILED DESCRIPTION:
A Phase 2 two-armed placebo-controlled, double-blind, randomized (1:1), multiple dose, single center interventional study to evaluate the safety and proof of concept for an antimicrobial decapeptide KSL-W chewing gum formulation 3 times per day over 4 treatment days measuring dental plaque regrowth from specific regions of the upper jaw, lower jaw, buccal and lingual surfaces.

ELIGIBILITY:
Inclusion Criteria:

* A negative urine pregnancy test (females of childbearing potential only)
* A negative urine drug test
* On a reliable form of birth control for at least 30 days prior to the start of the study and willing to use a reliable form of contraception for the duration of the study (Females of childbearing potential only), with reliable contraception defined as:
* Abstinence which has been the customary lifestyle of choice
* Oral contraceptive, either estrogen progesterone combined, or progesterone alone
* Injectable progesterone
* Implants of levonorgestrel
* Estrogenic vaginal ring
* Percutaneous contraceptive patches
* Intrauterine device or intrauterine system
* Double barrier method [condom or occlusive cap (diaphragm or cervical vault caps) plus spermicidal agent (foam, gel, film, cream, suppository)]
* Male partner sterilization at least 6 months prior to the female subject's entry into the study, and this male is the sole partner for that subject
* Post-menopausal for at least two years
* Good health, as determined by pertinent medical history, physical examination, and vital signs
* A minimum of 20 natural teeth with 6 scorable surfaces per tooth
* Sufficient number of opposing posterior teeth to chew on both sides of the mouth as determined by the examining dentist
* Teeth that have gross caries, full crowns or extensive restorations on facial and/or lingual surfaces, orthodontic bands, and third molars are not included in the tooth count
* Subject must have refrained from all oral hygiene procedures 12 to 16 hours prior to screening visit
* Plaque Index of 1.95 or greater (Turesky et al-1970)
* Willing to forgo any optional dental procedures during the study period, such as dental prophylaxis or teeth whitening
* Ability to comprehend and a willingness to sign an informed consent, which includes the Authorization for the Release of Health Information document
* Ability to access the internet to complete the drug compliance information
* Willingness to comply with all study procedures

Exclusion Criteria:

E01 Phenylketonuria E02 Acute or chronic medical conditions, organ system disease, or medications that, in the principal investigator's opinion, would impair the subject's ability to participate E03 TMD E04 Self-reported allergy to sucralose or mint flavors E05 Self-reported use of tobacco products including e-cigarettes E06 Use of any type of anticoagulant medications (eg clopidogrel) E07 Routine use of proton pump inhibitors E08 Allergic to any component of the study drug E09 Gross oral pathology, including widespread caries or chronic neglect, extensive restoration, pre-existing gross plaque or calculus, or soft or hard tissue tumor of the oral cavity E010Orthodontic appliances or removable partial dentures that will compromise the ability of the potential subject to participate in the study E011Periodontitis as indicated by periodontal pockets greater than 4 millimeters on more than one site E012 Receipt of any investigational drug/test product within 30 days prior to study entry with study entry defined as Day 0, or currently participating in either the active or follow-up phase of any other investigational study or planning to participate in any other investigational study during participation in this trial E013 Participation in the Phase 1/2a antiplaque study E014 Receipt of antibiotics within 30 days prior to study entry E015 Need for antibiotic prophylaxis prior to invasive dental procedures E016 Receipt of prescription antibacterial oral products (eg products containing chlorhexidine) within 30 days prior to study entry E017 Pregnant or breast-feeding female E018 An employee of the study site directly involved with the study E019 Inability to comply with assigned treatment regimen

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery L Milleman, DDS, MPA, Principal Investigator — Salus Research

REFERENCES:
- [Derived] Kirkwood B, Miller M, Milleman J, Milleman K, Leung K. Four-day plaque regrowth evaluation of a peptide chewing gum in a double-blind randomized clinical trial. Clin Exp Dent Res. 2020 Jun;6(3):318-327. doi: 10.1002/cre2.275. Epub 2019 Dec 14. PMID 32558314

RESULTS

PARTICIPANT FLOW:
Groups:
- KSL-W 30 mg: 3 times per day over 4 treatment days
  KSL-W: Plaque reducing gum
- Chewing Gum Placebo: 3 times per day over 4 treatment days
  Chewing Gum Placebo
Period: Overall Study
Arm/Group | KSL-W 30 mg | Chewing Gum Placebo
Started | 14 | 13
Completed | 13 | 13
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KSL-W 30 mg | Chewing Gum Placebo | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 11 | 13 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 13 | 23
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety, Tolerability and Effectiveness in Reducing Dental Plaque of KLS-W Delivered in a Chewing Gum Formulation
Description: Day 4 Exam Following 72-hours of Chewing Gum Treatment. Exam Included Vital Signs and Whole Mouth Dental Examination (Maxillary Buccal, Maxillary Lingual, Mandibular Buccal and Mandibular Surfaces) Assessing for Local Oral Mucosal Reactions, Systemic Reactions and Serious Total Body Reactions.
Time Frame: Baseline, and Day 4 Following Three-days of Chewing Gum Treatment
Population: 26 Male and female subjects undergoing exam following 72-hours of Chewing Gum Treatment with results compared to baseline
Measure: Number; unit: participants
Groups:
- Chewing Gum Placebo: 3 times per day over 4 treatment days
  Placedo Chewing Gum
Arm/Group | KSL-W 30 mg | Chewing Gum Placebo
Number analyzed (Participants) | 13 | 13
participants
  Local Oral Mucosal Changes | 0 | 0
  Systemic Reactions or Serious Total Body Reactions | 0 | 0

2. Secondary Outcome: Score on a Scale of Whole Mouth Change in Plaque Regrowth Based on Sub-scores From Specific Regions of the Upper Jaw, Lower Jaw, Buccal and Lingual Surface Using Standardized QHT Measures
Description: The Amount of Plaque Regrowth Based on Sub-scores From Specific Regions of the Upper Jaw, Lower Jaw, Buccal and Lingual Surface Based on the Quigley-Hein Turskey Plaque Index (QHT) a measure that evaluates plaque on teeth surfaces on a scale of 0 to 5 defined by Quigley &Hein in 1962 and modified by Turskey et al in 1970. All teeth except the third molars are assessed. An index for the entire mouth is determined by dividing the total score by the number of surfaces examined. Quigley-Hein-Turskey Plaque Index Scale Minimum score 0=no plaque, 1-Isolated flecks of plaque at the gingival margin, 2=A continuous band of plaque up to 1mm at the gingival margin, 3=Plaque greater than 1mm in width and covering up to one third of the tooth surface, 4=Plaque covering from one thirds to two thirds of the tooth surface, Maximum score of 5=Plaque covering more than two thirds of the tooth surface
Time Frame: 4 Days
Population: Summary of Quigley-Hein-Turskey Plaque Index Scores, Whole Mouth and by Quadrants baseline (Day 0) and day following 72-hours of treatment (Chewing gum 3x/day)
Measure: Mean (Standard Deviation); unit: QHT Score, Subscore
Groups:
- KSL-W 30 mg: 3 times per day over 4 treatment days (Day 0)
  KSL-W: Plaque reducing gum
Arm/Group | Chewing Gum Placebo | KSL-W 30 mg
Number analyzed (Participants) | 13 | 13
QHT Score, Subscore
  Whole Mouth Quigley-Hein-Turskey Plaque Score (Day 0) | 2.95 (0.471) | 2.96 (0.403)
  Maxillary Buccal Quigley-Hein-Turskey Plaque Score (Day 0) | 3.05 (0.712) | 2.96 (0.576)
  Maxillary Lingual Quigley-Hein-Turskey Plaque Score (Day 0) | 2.52 (0.572) | 2.49 (0.434)
  Mandibular Buccal Quigley-Hein-Turskey Plaque Score (Day 0) | 3.07 (0.513) | 2.80 (0.550)
  Mandibular Lingual Quigley-Hein-Turskey Plaque Score (Day 0) | 3.20 (0.676) | 3.60 (0.663)
  Whole Mouth Quigley-Hein-Turskey Plaque Score (Day 4) | 2.80 (0.680) | 1.65 (0.725)
  Maxillary Buccal Quigley-Hein-Turskey Plaque Score (Day 4) | 3.63 (0.679) | 2.85 (1.064)
  Maxillary Lingual Quigley-Hein-Turskey Plaque Score (Day 4) | 1.81 (0.558) | 0.50 (0.477)
  Mandibular Buccal Quigley-Hein-Turskey Plaque Score (Day 4) | 3.23 (0.945) | 2.16 (1.011)
  Mandibullar Lingual Quigley-Hein-Turskey Plaque Score (Day 4) | 2.52 (0.858) | 1.14 (0.779)

ADVERSE EVENTS:
Time Frame: 30 mg KSL-W administered in a chewing gum formulation 3 times per day over 4 treatment days. Oral hygiene (teeth brushing, flossing and/or mouth wash rinse) was prohibited throughout the trial, beginning 12 to 16 hours before both the screening and Baseline (Day 0) visits, during the 4 days of treatment (Days 0, 1, 2, and 3), and ending after the periodontal examination and plaque assessment on Day 4.
Description: Any AE that occurred after administration of the first dose of study treatment or any medical or dental condition present at baseline but worsened in intensity. Including AE incidence rates by system organ class (SOC) and by preferred term (PT) within SOC. Incidence rates as number of treatment emergent AEs divided by the total number of patient-weeks. AE incidence proportion is the number of subjects having at least one AE of a particular type divided by the number of subjects exposed
Arm/Group | KSL-W 30 mg | Chewing Gum Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT02864901/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT02864901/SAP_001.pdf
  • Informed Consent Form (2016-06-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT02864901/ICF_002.pdf